CLINICAL TRIAL: NCT06418048
Title: Prospective Registry and Biobank of Patients With Infectious Diseases
Brief Title: INfectious DIsease REgistry BIObank
Acronym: INDI-REBIO
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Castagna Antonella, Full Professor, Ospedale San Raffaele
Other Study IDs: CET 138-2023
Record Dates: First submitted 2024-01-31; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Bloodstream Infections; Central Nervous System Infections; Bone and Joint Infections; Endovascular Infections; Infective Endocarditis; CIED-related Infections; Vertebral Osteomyelitis
MeSH Terms: conditions — Sepsis; Central Nervous System Infections; Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — * Blood
  * Cerebrospinal fluid (CSF)
  * Respiratory specimens
  * Synovial fluid
  * Urine
  * Stool
  * Seminal fluid
  * Tissue samples
  * Microbial isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study designed to describe the clinical, laboratory, imaging, microbiological characteristics and treatment of specific infectious diseases, with the addition of a dedicated biobank.

DETAILED DESCRIPTION:
The registry would provide a comprehensive database including a vast population of patients with infectious diseases, favoring the analysis of clinical, laboratory and therapeutic data of specific infectious conditions.

Specific infectious diseases of major interest include, among others:

* Bloodstream infections (i.e.: infectious syndromes manifesting with bacteremia)
* Endovascular infections (i.e.: infective endocarditis, cardiovascular implantable electronic device infections, vascular graft infections, etc.)
* Central nervous system infections (i.e.: meningitis, encephalitis, cerebral abscess, ventricular shunts infections, etc.)
* Bone and joint infections (i.e.: osteomyelitis, spondylodiscitis, prosthetic joint infections, etc.)
* Sexually transmitted infections (i.e.: gonococcal and non-gonococcal urethritis, proctitis, epididymo-orchitis, syphilis, etc.)
* HIV infection
* Emerging and re-emerging infectious diseases.

General objectives of the study for each specific infectious disease include:

* description and evolution over time of clinical and laboratory characteristics of patients with specific infectious diseases;
* description and evolution over time of microbial isolates, including antimicrobial susceptibility testing;
* description and evolution over time of treatment employed in patients with specific infectious diseases;
* evaluation of predictive factors for treatment success and mortality in patients with specific infectious diseases;
* description, evaluation and prognostic impact of microbial, immunological and inflammatory biomarkers.

The general study objectives, along with more specific objectives related to a specific infectious disease, will be evaluated in specific observational studies, nested within the Registry (i.e., using data and biosamples collected in the Registry with the potential addition of data obtained from investigations performed on available biological samples).

To achieve these objectives, participants are asked to donate biological samples (blood, cerebrospinal fluid, urine, other relevant biological samples related to the specific infectious disease, collected according to good clinical practice and available guidelines) for studies to identify modifiers of a specific infectious disease and to establish and validate biological markers tracking the progressive course of the considered disease, along with drug efficacy and toxicity.

The following clinical and laboratory data will be recorded at baseline and at follow-up visits:

* Age, measured in years
* Sex at birth (male, female)
* Comorbidities, measured with Charlson score (minimum 0 - maximum 37; higher scores linked to worse outcome)
* Source of infection, (central nervous system, respiratory tract, endovascular infection, intra-abdominal, urinary tract, skin and soft tissue, bone and joint, other).
* Sequential Organ Failure Assessment (SOFA) score (minimum 0 - maximum 24; higher scores linked to worse outcome)
* Pitt Score (minum 0 - maximum 14; higher scores linked to worse outcome)
* Length of hospital stay (days)
* Number of patients requiring Intensive care unit (ICU) admission, surgical interventions or other procedures
* Nerological impairment (Rankin scale [minimum 0 - maximum 6; higher scores linked to worse outcome])
* Functional impairment (Karnofsky scale [minum 0 - maximum 100; higher scores linked to better outcome])
* Results of routine laboratory tests
* Drug plasma concentrations
* Results of microbiological investigations (identification of the causative organisms, antimicrobial susceptibility testing results, mechanism of resistance)
* Results of imaging investigations
* Treatment strategies (type, dose, administration of antimicrobials)
* Development of drug toxicities
* Mortality (all-cause and infection-attributable)

Both data and biosamples will be collected starting from the baseline (BL) of the infectious disease after obtaining informed consent. Follow-up data and biosamples will be collected at the end of treatment (EOT) and at 6 months after the EOT for the specific condition or, in case of no therapeutic intervention, at 6 months after diagnosis. In patients with HIV infection follow-up data and biosamples will be collected yearly after baseline. Additional data and biosamples will be collected at other time-points according to the usual temporal evolution of specific diseases, and in case of relevant clinical events or therapeutic modification. All specimens will be collected according to good clinical practice and available national and international guidelines.

Data analysis will be performed by the investigators on approved proposals. Statistical methods will be defined as part of the proposals.

The variables of the study will be described using means or medians and 95% confidence intervals or interquartile ranges for continuous variables and proportions with their 95% confidence intervals for categorical variables.

Comparisons between groups will be made using the chi-square test or Fisher's exact test (categorical variables) or using the non-parametric Mann-Whitney test (continuous variables).

Significant variations in continuous variables over time may be assessed using t-tests for paired data o Wilcoxon ranks sign test (only two timepoints) o analysis of variance for repeated measures or linear mixed models (all timepoints available during follow-up).

The presence of linear relationships between continuous variables can be tested by means of Pearson correlation coefficients (parametric) or Spearman correlation coefficients (non-parametric).

Logistic regression models will be applied to determine the predictors of outcomes; the risks (odds ratios) and the corresponding 95% confidence intervals will be reported.

Cox regression models will be applied to determine predictors of outcomes; risks (odds ratios) and corresponding 95% confidence intervals will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected or microbiologically documented infectious diseases (bacterial, viral, fungal or parasitic);
* At least 18 years of age or older;
* Able to provide informed consent;
* Participants who are unable to understand the study protocol or are unable to give informed consent, but have a legal representative

Exclusion Criteria:

- Participants who are unable to understand the study protocol or are unable to give informed consent, and have no legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with specific infectious diseases followed at the IRCCS San Raffaele Hospital (either as inpatients or outpatients).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2044-01-31 (Estimated); Study Completion 2044-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of specific infectious diseases | 6 months (with the exception of people living with HIV)
  Describe the clinical presentation of specific infectious diseases, by means of Sequential Organ Failure Assessment (SOFA) score (minimum 0 - maximum 24; higher scores linked to worse outcome).
Microbiological characteristics of specific infectious diseases | 6 months (with the exception of people living with HIV)
  Describe the microbiological characteristics of specific infectious diseases. Specifically:
  * Identification of the causative organisms
  * Antimicrobial susceptibility testing results
  * Mechanism of resistance
Treatment of specific infectious diseases | 6 months (with the exception of people living with HIV)
  Describe the antimicrobial treatment of specific infectious diseases

SECONDARY OUTCOMES:
Predictive factors of microbiological cure | 6 months (with the exception of people living with HIV)
  Describe the predictive factors of microbiological cure, defined as negativization of cultures from the infected site
Predictive factors of clinical cure | 6 months (with the exception of people living with HIV)
  Describe the predictive factors of clinical cure, defined as resolution of symptoms and signs attributable to the specific infectious disease
Need for surgical intervention or other procedures | 6 months (with the exception of people living with HIV)
  Describe the number of patients needing surgical intervention or other procedures
Need for ICU | 6 months (with the exception of people living with HIV)
  Describe the number of patients needing ICU transfer
Overall mortality | 6 months (with the exception of people living with HIV)
  Describe mortality due to any cause
Infection-attributable mortality | 6 months (with the exception of people living with HIV)
  Describe mortality due to the specific infectious disease
Neurological impairment | 6 months (with the exception of people living with HIV)
  Describe the extent of neurological impairment (Rankin scale [minimum 0 - maximum 6; higher scores linked to worse outcome])
Functional impairment | 6 months (with the exception of people living with HIV)
  Describe the extent of functional impairment (Karnofsky scale [minum 0 - maximum 100; higher scores linked to better outcome])
Development of comorbidities | 6 months (with the exception of people living with HIV)
  Describe the development of comorbidities (e.g. diabetes, cardiovascular diseases, etc.)
Development of drug toxicity | 6 months (with the exception of people living with HIV)
  Describe the development of drug toxicities. Specifically, but not limited to:
  * Nephrotoxicity, measured with serum creatinine levels (milligrams per deciliter)
  * Hepatotoxicity, measured with alanine aminotransferase and aspartate aminostrasferase (units per liter), bilirubin (milligrams per deciliter), prothrombin time (seconds)
  * Hematological Toxicity, measured with complete blood cell count (cells per microliter), hemoglobin (grams per deciliter), platelets (count per microliter)
  * Cardiotoxicity, evaluated with electrocardiogram monitoring for arrhythmias
  * Neurotoxicity, measured with Rankin scale (minimum 0 - maximum 6; higher scores linked to worse outcome)
  * Gastrointestinal Toxicity, measured with Bristol stool chart

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ripa, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ripa M, Galli L, Cinque P, Nozza S, Spagnuolo V, Tassan Din C, Guffanti M, Lolatto R, Piromalli G, Carletti S, Locatelli M, Sanvito F, Ponzoni M, Cantarelli E, Tresoldi C, Castagna A; INDI-REBIO Study Group. The INfectious DIsease REgistry BIObank (INDI-REBIO): protocol for the design and implementation of a single-centre, prospective registry and biobank in a tertiary care centre in Italy for advancing infectious disease research. BMJ Open. 2025 Aug 12;15(8):e091113. doi: 10.1136/bmjopen-2024-091113. PMID 40803735